CLINICAL TRIAL: NCT05712265
Title: A Phase 1, Open-Label, Fixed-Sequence Crossover Study to Evaluate the Effect of a Strong Inhibitor of Cytochrome P450 2C19 on the Pharmacokinetics of Miricorilant in Healthy Subjects
Brief Title: Study to Evaluate the Effects of a Cytochrome P450 2C19 Inhibitor on the Pharmacokinetics of Miricorilant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT118335-856
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Antipsychotic Induced Weight Gain; Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — CORT118335; Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Miricorilant - Fluvoxamine/Miricorilant (Experimental): Participants will receive a single oral dose of miricorilant 600 mg on Days 1 and 10 and a single oral dose of fluvoxamine 50 mg on Days 4 to 12.
  Interventions: Drug: Miricorilant; Drug: Fluvoxamine

INTERVENTIONS:
Drug: Miricorilant — Miricorilant 6 x 100 mg coated tablets
  Other Names: CORT118335
Drug: Fluvoxamine — Fluvoxamine 50 mg tablet

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of miricorilant in the presence and absence of the strong cytochrome P450 [(CYP) 2C19] inhibitor, fluvoxamine, in healthy participants. Participants will receive a single dose of miricorilant under fed conditions with a standard breakfast after an overnight fast alone and in combination with once-daily doses of fluvoxamine. Blood samples will be collected at regular intervals for PK and safety analysis between admission and discharge from the clinical unit.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand a written informed consent
* Willing and able to comply with all study requirements including potential CYP 2C19 genotyping analysis
* Male participants must agree to use an adequate method of contraception
* Healthy men or non-pregnant, non-lactating healthy women of non-childbearing potential
* Body mass index of 19.0 to 32.0 kg/m^2
* Body weight ≥50 kg.

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment. Hay fever is allowed unless it is active.
* Significant skin disease, including rash, food allergy, eczema, psoriasis, or urticaria
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease (except cholecystectomy), bleeding disorder, neurological or psychiatric disorder, as judged by the Investigator
* Poor venous access that limits phlebotomy
* Evidence of current SARS-CoV-2 infection
* Clinically significant abnormal clinical chemistry, hematology, or urinalysis as judged by the Investigator. Participants with Gilbert's Syndrome are allowed.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* Evidence of renal impairment at screening
* Positive highly sensitive serum pregnancy test at screening or admission. Those who are pregnant or lactating will be excluded. A woman is considered of childbearing potential unless she is permanently sterile or is postmenopausal.
* Clinically-significant ECG abnormalities or vital sign abnormalities at screening or at baseline
* Have received any study drug in a clinical research study within 30 days (or 5 half-lives if longer) prior to first dose of study medication
* Are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 2 g per day acetaminophen or COVID-19 vaccines) in the 14 days before study drug administration. Exceptions may apply.
* Are currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months, or 3 months for inhaled products
* Are taking, or have taken, selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors within 3 months before study drug administration
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in men >21 units per week and women >14 units per week (1 unit = 12 oz 1 bottle/can of beer, 1 oz 40% spirit, or 5 oz glass of wine)
* Confirmed positive alcohol urine test at screening or admission
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Positive drugs of abuse test result
* Male participants with pregnant or lactating partners
* Donation of blood within 2 months or donation of plasma within 7 days prior to first dose of study medication
* Are, or are immediate family members of a study site or Sponsor employee
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of miricorilant (Cmax) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Days 1 and 10
Area under the curve from time zero to the time of last measurable plasma concentration of miricorilant (AUC0-last) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Days 1 and 10
Area under the curve from time zero extrapolated to infinity of plasma concentration of miricorilant (AUC0-inf) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Days 1 and 10

SECONDARY OUTCOMES:
Number of participants with one or more treatment-emergent adverse events (TEAEs) | Up to 30 days after study drug administration
Number of participants with one or more serious adverse events (SAEs) | Up to 30 days after study drug administration
Number of participants with a clinically-significant vital sign abnormality | Up to Day 13
Number of participants with a clinically-significant laboratory test abnormality | Up to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, PhD, Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No